CLINICAL TRIAL: NCT04085783
Title: PRP in Recurrent Implantation Failure , Hope or Hype
Brief Title: PRP in Recurrent Implantation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kamal Rageh (Other)
Responsible Party: Sponsor-Investigator, Dr. Kamal Rageh, medical director, Al Baraka Fertility Hospital
Organization: Al Baraka Fertility Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlBarakaBH
Record Dates: First submitted 2018-11-04; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Implantation Failure
Keywords: Recurrent implantation failure; implantation; IVF; platelet rich plasma (PRP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endometrial PRP (Experimental): In study group (75 patients), intrauterine infusion of PRP was done 48 hrs. before ET. PRP was prepared from autologous blood and it was made by using two steps centrifuge process. All Blastocyst transfers were performed under ultrasound guidance by one expert gynecologist with infertility fellowship. ET was performed according to American Society for Reproductive Medicine (ASRM) guidelines 2013 (Two or three embryos for each participant). On PRP infusion day, 17.5 ml of peripheral venous blood was drawn into a syringe that contains 2.5 ml of Acid Citrate and centrifuged immediately at 1200 rpm for 12 min to separate red blood cells, then plasma was centrifuged again at 3300 rpm for 7 min to obtain PRP that contained platelet 4-5 times more than peripheral blood. 0.5- 1 ml of PRP was infused into the uterine cavity with embryo transfer catheter (Wallace - Smiths, UK). On the other side, No PRP was done in control group. Pregnancy tests were done 12 days after ET.
  Interventions: Procedure: PRP

INTERVENTIONS:
Procedure: PRP — Platelet Rich Plasma

SUMMARY:
The endometrial function and endometrial receptivity have been accepted to be major limiting factors in the establishment of pregnancy. In spite of improved almost all aspects of IVF: ovarian stimulation, embryo culture and transfer, the pregnancy rates still not satisfactory. The bottleneck is the process of implantation.

Recurrent implantation failure (RIF) is one of the nightmares in reproductive medicine and despite several strategies that have been described for management; there is no universal agreement yet.

Recently, intrauterine infusion of platelet-rich plasma (PRP) is described to promote endometrial growth and receptivity, PRP has been investigated as a therapeutic approach for several medical disorders in dermatology and rheumatology, but its use in IVF is still limited.

Objective:

To evaluate the effectiveness of intrauterine perfusion of autologous platelet-rich plasma in the improvement of pregnancy rate in RIF patients.

DETAILED DESCRIPTION:
After ethical committee approval was obtained, 150 infertile women with history of RIF gave their written consent to be included in this study. All were recruited from the outpatient clinic of Al-Baraka fertility hospital - with age below 40 yrs, body mass index (BMI) below 30 kg/m2, whose uteri were morphologically normal as confirmed by HSG and U/S to limit additional factors that may affect the results of the study - Divided into 2 comparable groups; all participants underwent antagonist protocol, oocytes retrieval, fertilization and embryo transfer; In the study group, intrauterine infusion of 0.5 to 1 ml of platelet-rich plasma (PRP) was performed 48 hrs before blastocyst transfer, pregnancy tests were done 12 days after ET.

ELIGIBILITY:
Inclusion Criteria:

* female infertile patients with history of recurrent implantation failure
* age below 40 yrs.,
* body mass index (BMI) below 30 kg/m2.

Exclusion Criteria:

* haematological and immunological disorders
* hormonal disorders,
* chromosomal and genetic abnormalities and uterine abnormalities (acquired or congenital) as confirmed by HSG and U/S to limit additional factors that may affect the results of the study

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-12-03 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with positive pregnancy test | 2 weeks
  B-hCG ; pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Al-BARAKA FERTILITY HOSPITAL, Manama, Adliya, Bahrain